CLINICAL TRIAL: NCT03608865
Title: Phase II Trial of Durvalumab (MEDI4736) and Tremelimumab in Hormone Receptor-positive, Hypermutated Metastatic Breast Cancer Identified by Whole Exome Sequencing
Brief Title: Durvalumab (MEDI4736) and Tremelimumab in Hormone Receptor-positive, Hypermutated Metastatic Breast Cancer Identified by Whole Exome Sequencing
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2016-0912
Record Dates: First submitted 2018-07-23; First posted 2018-08-01 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Intervention Model Description: Drug:Durvalumab + tremelimumab Dose/Potency: Durvalumab 1500mg(up to 4cycle) / tremelimumab 75mg(up to 13 cycle) Dose Frequency:Q4W Route of Administration:IV infusion Regimen/Treatment Period:Day 1 of each 4 week cycle Use:Experimental
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): Drug:Durvalumab + tremelimumab Dose/Potency:Durvalumab 1500mg(up to 4cycle) / tremelimumab 75mg(up to 13 cycle) Dose Frequency:Q4W Route of Administration:IV infusion Regimen/Treatment Period:Day 1 of each 4 week cycle Use:Experimental
  Interventions: Drug: Durvalumab with Tremelimumab

INTERVENTIONS:
Drug: Durvalumab with Tremelimumab — Trial treatment should be administered on Day 1 of each cycle after all procedures/assessments have been completed as detailed on the Trial Flow Chart. Trial treatment may be administered up to 3 days before or after the scheduled Day 1 of each cycle due to administrative reasons. All trial treatments will be administered on an outpatient basis. Durvalumab 1500mg + tremelimumab 750 mg will be administered as a 60 minute each one IV infusion every 4 weeks. Sites should make every effort to target infusion timing to be as close to 60 minutes as possible. However, given the variability of infusion pumps from site to site.

SUMMARY:
Abbreviated Title : Durvalumab + tremelimumab in hypermutated breast cancer Trial Phase : II Clinical Indication : Hormone receptor-positive metastatic breast cancer Trial Type : Interventional Type of control : None Route of administration : Intravenous Trial Blinding : None Treatment Groups : Durvalumab + tremelimumab Number of trial subjects : Approximately 150 patients will be prescreened with whole exome sequencing. Then 30 patients will be enrolled in the treatment phase.

Estimated enrollment period : 24 months Estimated duration of trial : The sponsor estimates that the trial will require approximately 48 months from the time the first subject signs the informed consent until the last subject's last visit.

Duration of Participation : 24 months Estimated average length of treatment per patient : 8 months

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
* Pre or postmenopausal women with stage IV hormone receptor-positive breast cancer by histological or cytological confirmation
* Age > 19 years at time of study entry
* Progression after one line of any systemic therapy (endocrine, targeted or chemotherapy) in the metastatic setting
* 2.1 or more nonsynonymous mutations per megabase (Mb) by WES
* Subject who has biopsy-accessible tumor
* At least one measurable lesion by RECIST 1.1. Biopsied tumor may be counted a measurable lesion if it is not excised
* Documented disease progression on the most recent therapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 ~ 1
* Life expectancy of > 12 weeks
* Adequate normal organ and marrow function as defined below:

  1. Haemoglobin ≥ 9.0 g/dL
  2. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (> 1500 per mm3)
  3. Platelet count ≥ 100 x 109/L (>100,000 per mm3)
  4. Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN). This will not apply to subjects with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
  5. AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤ 5x ULN
  6. Serum creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance: ① Males: Creatinine CL (mL/min) = Weight (kg) x (140 - Age) 72 x serum creatinine (mg/dL), ② Females: Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL)
* Female subjects must either be of non-reproductive potential (ie, post-menopausal by history: ≥ 60 years old and no menses for 1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry. Otherwise, subjects must adhere to acceptable forms of birth control (a physician-approved contraceptive method: oral, injectable, or implantable hormonal contraceptive; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner).
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site). Previous enrollment in the present study
* Participation in another clinical study with an investigational product during the last 4 weeks
* Any previous treatment with a PD-1 or PD-L1 inhibitor, including durvalumab or an anti-CTLA-4, including tremelimumab
* Previous or coexisting malignancies. However, malignancies that have been curatively treated >5 years prior to study entry can be included. Exceptionally, cervical cancer in-situ, basal cell carcinoma, papillary thyroid carcinoma and superficial bladder tumors (T1a and Tis) can be included anytime after curative treatment
* Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) ≤ 21 days prior to the first dose of study drug and within 6 weeks for nitrosourea or mitomycin C) for sufficient wash-out time
* Palliative radiation, whole brain radiotherapy (WBRT), or gamma knife surgery (GKS) for brain metastases ≤ 2 weeks prior to initiation of study medication. Major surgery ≤ 4 weeks or minor surgery ≤ 2 weeks prior to initiation of study medication. Majority or minority of surgery can be decided at the investigator's discretion. Subjects who received these local therapy may be enrolled after predetermined time period
* Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Fredericia's Correction
* Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab or tremelimumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid
* Any unresolved toxicity (≥CTCAE grade 2) from previous anti-cancer therapy. Subjects with irreversible toxicity that is not reasonably expected to be exacerbated by the investigational product may be included (e.g., hearing loss, peripherally neuropathy)
* Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE >Grade 1
* Active or prior documented autoimmune disease within the past 2 years NOTE: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
* Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
* History of primary immunodeficiency
* History of allogeneic organ transplant
* History of hypersensitivity to durvalumab or tremelimumab
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have evidence of acute or chronic hepatitis A (anti-HAV antibody+), hepatitis B (HBs antigen+), hepatitis C (anti-HCV antibody+) or human immunodeficiency virus (HIV-1 or HIV-2 antibody+ or HTLV-1 antibody+), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
* Known history of previous clinical diagnosis of tuberculosis
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab or tremelimumab
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
* Symptomatic brain metastasis or leptomeningeal seeding. However, after WBRT or GKS for symptomatic brain or leptomeningeal metastases, if subjects are stable for 4 weeks without steroid and the dosage of anti-convulsant is stable for 4 weeks, they are eligible. Asymptomatic central nervous system metastases are eligible if the subject has no abnormal findings on neurologic examination and is not receiving corticosteroid therapy to control symptoms
* Subjects with uncontrolled seizures
* Female patients who are pregnant or breastfeeding or female subjects of reproductive potential who are not willing to employ effective birth control from screening to 180 days after the last dose of durvalumab + tremelimumab combination therapy or 90 days after the last dose of durvalumab monotherapy, whichever is the longer time period

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pre or postmenopausal women with stage IV hormone receptor-positive breast cancer by histological or cytological confirmation
Enrollment: 30 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) by RECIST 1.1 | up to 4 years (the end of study)
  To evaluate objective response rate (ORR) based on RECIST 1.1 in hormone receptor-positive, hypermutated metastatic breast cancer identified by whole exome sequencing (WES) Hypothesis: Durvalumab + tremelimumab in patients with hormone receptor-positive, hypermutated metastatic breast cancer identified by WES will result in clinically meaningful ORR based on RECIST 1.1

SECONDARY OUTCOMES:
Clinical benefit rate (CBR) by RECIST 1.1 defined by complete or partial response or stable disease for at least 24 weeks | every 1 year up to 4 years (the end of study)
  To evaluate clinical benefit rate (CBR) by RECIST 1.1 defined by complete or partial response or stable disease for at least 24 weeks
Duration of response (DoR) | every 1 year up to 4 years (the end of study)
  To evaluate duration of response (DoR)
Disease control rate (DCR) by RECIST 1.1 | every 1 year up to 4 years (the end of study)
  To evaluate disease control rate (DCR) by RECIST 1.1
Progression-free survival (PFS) by RECIST 1.1 | every 1 year up to 4 years (the end of study)
  To evaluate progression-free survival (PFS) by RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei Cancer Center, Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No